CLINICAL TRIAL: NCT00997321
Title: Propofol Versus Ketamine for Procedural Sedation During Painful Procedures in the Emergency Department
Brief Title: Propofol Versus Ketamine for Moderate Procedural Sedation in the Emergency Department (ED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMRF062661
Record Dates: First submitted 2009-10-12; First posted 2009-10-19 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Sedation
Keywords: ketamine; propofol; procedural sedation; moderate procedural sedation in the ED
MeSH Terms: interventions — Propofol; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Active Comparator): propofol 1 milligram per kilogram intravenous bolus followed by 0.5 millligrams per kilogram as needed for mooderate procedural sedation
  Interventions: Drug: propofol
- Ketamine (Active Comparator): ketamine 1 milligram per kilogram followed by 0.5 millgram per kilogram as needed for moderate procedural sedation
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: propofol — propofol 1 millgram per kilogram intravenous bolus followed by 0.5 milligrams per kilogram as needed for moderate procedural sedation
  Arms: Propofol
Drug: Ketamine — ketamine milligram per kilogram followed by 0.5 milligrams per kilogram as need for moderate procedural sedation
  Arms: Ketamine

SUMMARY:
This study is a clinical trial of moderate sedation with propofol versus moderate sedation with ketamine for procedural sedation in the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* patients who require moderate procedural sedation with propofol in the ED

Exclusion Criteria:

* age > 17 years
* pregnant
* intoxicated
* cannot give informed consent
* allergy to ketamine or propofol
* patient will require deep procedural sedation
* ASA physical status score > 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Miner, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Miner JR, Gray RO, Bahr J, Patel R, McGill JW. Randomized clinical trial of propofol versus ketamine for procedural sedation in the emergency department. Acad Emerg Med. 2010 Jun;17(6):604-11. doi: 10.1111/j.1553-2712.2010.00776.x. PMID 20624140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 patients recruited in the Emergency Department
Pre-assignment Details: 97 enrolled subjects underwent procedural sedation
Groups:
- Propofol: propofol 1 milligram per kilogram at the start of the procedure followed by 0.5 milligrams per kilogram every 3 minutes as needed for moderate procedural sedation
- Ketamine: ketamine 1 milligram per kilogram intravenous bolus to start procedure followed by 0.5 mg/kg every three minutes as needed for moderate procedural sedation
Period: Overall Study
Arm/Group | Propofol | Ketamine
Started | 50 | 50
Completed | 50 | 47
Not Completed | 0 | 3
Not completed — did not undergo sedation after enrollmen | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol | Ketamine | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34 (5) | 30 (5) | 32 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 26 | 25 | 51
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Depression (Sub-clinical and Clinical Signs)
Description: binary measure based on the occurrence of an oxygen saturation less than 93 at any time, a change in baseline end tidal co2 >10 or an absence on capnographic waveform
Time Frame: From one minute prior to start of the procedure until the patient has returned to baseline mental status after the conclusion of the sedation procedure up to 60 minutes)
Population: 50 subjects were randomized to each group, 50 subjects in the propofol arm completed the study, 47 in the ketamine arm
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Propofol; Ketamine: percentage of participants with respiratory depression
Arm/Group | Propofol | Ketamine
Number analyzed (Participants) | 50 | 47
percentage of participants | 0.4 [0.26 to 0.55] | 0.6 [0.45 to 0.74]

2. Secondary Outcome: Time to Return of Baseline Mental Status
Description: time in seconds from the first dose of medication until the patient has regained baseline mental status
Time Frame: from start of procedure until the return of baseline mental status up to 120 minutes
Population: 50 patients were randomized to the propofol group and 50 to ketamine, 50 underwent the procedure in the propofol group and 47 in the ketamine group
Measure: Median (95% Confidence Interval); unit: minutes
Groups:
- Propofol; Ketamine: time in minutes from the start of the procedure until the return of baseline mental status
Arm/Group | Propofol | Ketamine
Number analyzed (Participants) | 50 | 47
minutes | 5 [4 to 6] | 14 [10 to 29]

3. Secondary Outcome: Patient Reported Pain or Recall of the Procedure
Description: patient completed question after return to baseline mental status "did you feel pain during the procedure" and "do you remember any part of the procedure" answered by circling yes or no on a question sheet, positive if yes to either question
Time Frame: single measurement immediately after patient returns to baseline mental status after sedation procedure
Population: 100 patients were randomized, 50 to each group, 50 underwent the procedure in the propofol group and 47 in the ketamine group
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Propofol: percentage of subjects reporting pain after the procedure who received propofol
- Ketamine: percentage of subjects reporting pain after the procedure who received ketamine
Arm/Group | Propofol | Ketamine
Number analyzed (Participants) | 50 | 47
percentage of participants | 0.06 [0.01 to 0.17] | 0.02 [0.001 to 0.11]

4. Secondary Outcome: Depth of Sedation
Description: Observes assesment of alertness scale, 1-5 ordinal scale measuring level of awareness, one represents awake, 5 general anesthesia/unresponsive to pain
Time Frame: single measurement during sedation procedure
Population: 100 patients were randomized, 50 to the propofol group, 50 of whom underwent sedation, and 50 in the ketamine group, 47 of whom underwent sedation
Measure: Median (Full Range); unit: score on a scale
Groups:
- Propofol: median depth of sedation by the observers assesment of alertness scale in the propofol group
- Ketamine: median depth of sedation by the observers assesment of alertness scale in the ketamine group
Arm/Group | Propofol | Ketamine
Number analyzed (Participants) | 50 | 47
score on a scale | 2 [1 to 4] | 2 [1 to 4]

ADVERSE EVENTS:
Arm/Group | Propofol | Ketamine
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/47
Other Adverse Events (participants affected / at risk) | 0/50 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No